CLINICAL TRIAL: NCT06299670
Title: Efficacy of Combination of Hdroxyurea and Thalidomide Over Either Hydroxyurea or Thalidomide Alone in the Treatment of Transfusion Dependent Thalassemia in Children: A Quasi-Randomised Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, MD ANWARUL KARIM, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 939
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Transfusion-dependent Thalassemia
Keywords: Trnafusion dependent thalssemia, Hydroxyurea, Thalidomide
MeSH Terms: interventions — Thalidomide; Hydroxyurea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thalidomide (Experimental): Patient getting Thalidomide
  Interventions: Drug: Thalidomide
- Hydroxyurea (Experimental): Hydroxyurea
  Interventions: Drug: Hydroxy Urea
- Combination (Experimental): combination of Thalidomide & Hydroxyurea
  Interventions: Drug: Combinations

INTERVENTIONS:
Drug: Thalidomide — Patients will get only Thalidomide
  Arms: Thalidomide
Drug: Hydroxy Urea — Patients will get only Hydroxyurea
  Arms: Hydroxyurea
Drug: Combinations — Combination Of Thalidomide & Hydroxyurea
  Arms: Combination

SUMMARY:
Transfusion Dependent Thalassemia (TDT) is an emerging global public health concern. Hemopoietic stem cell transplantation (HSCT) is the only curative treatment. But its adoption is limited due to lack of HLA matched donor, experienced centers and high initial cost. So, researches are going on in search of an effective, safe, easily available treatment option. Use of fetal haemoglobin inducing agents shows promising effects in treatment of TDT patients. Thalidomide an immunomodulating and anti-angiogenic drug has been shown to induce γ-globin gene expression and increase the proliferation of erythroid cells. Furthermore Hydroxyurea (HU) is known to increase haemoglobin (Hb) by HbF induction and reduction of inflammation and hypercoagulability.

Recent studies with combination of HU and Thalidomide have shown promising results in treatment of Thalassemia patients. However, most of those studies are retrospective or single arm nonrandomized trials & The study population includes both adult and children age group . So the effectiveness of combination therapy of Thalidomide and HU needs to be established through randomized trials.

This single centered non blinded quasi randomized clinical trial will be conducted at the Department of Pediatric Hematology and Oncology in Bangabandhu Sheikh Mujib Medical University (BSMMU), Bangladesh for one year of period. Thirty transfusion dependent thalassemia children of 3-18 years old will be included in each group. The objective of this study is to assess the effectiveness of combination of Thalidomide and Hydroxyurea in TDT children. It will play an important role in planning a cost effective and affordable treatment option for TDT children.This study will involve minimum physical risk to the patient. Written informed consent will be taken from parents or study subjects after brief explanation of the purpose and procedure. They will also be informed about the freedom to participate or not to participate at any time. Privacy and confidentiality will be safe guarded. History regarding age, sex, height, weight of these patients will be taken. Thorough physical examinations and laboratory investigations including CBC, Hb electrophoresis, serum Ferritin, serum creatinine, SGPT will be done. Data will be collected in a predesigned questionnaire and will be kept confidential. Statistical analysis will be done using the statistical software SPSS.

DETAILED DESCRIPTION:
Thalassemia is a monogenic hematological disorder caused as a result of defect in synthesis of globin chains of hemoglobin (Rachmilewitz et al., 2011; Cappellini et al., 2018). It causes ineffective erythropoiesis & lysis of red blood cells due to relative excess of unaffected globin chain (Rachmilewitz et al., 2011; Chen et al.,2021).

Annually about 50,000 children with a severe form of thalassemia (β-thalassemia major and HbE β-thalassemia) born globally among which 26,000 patients are regular blood transfusion dependent (Hossain et al, 2017; Cappellini et al., 2018; Shah et al, 2019). About 70-75% patients are found in southeast asia & eastern mediterranean region (Weatherall D.J., 2017).

Hematopoietic stem cell transplant (HSCT) is the only curative treatment option for homozygous thalassemia patients (Cappellini et al., 2018; Costa et al.,2022) . Unfortunately its application is limited due to scarcity of HLA-matched donor, high cost , lack of specialized dedicated centers and risk of transplant related morbidity and mortality (Cappellini et al., 2018; Shah et al, 2019; Lu et al.,2022).

Regular blood transfusion is an essential life saving supportive care to maintain growth and development in children with severe β-thalassemia (Cappellini et al., 2018; Shah et al, 2019; Ansari et al, 2022). However, Long term blood transfusion causes iron overload with cardiac, hepatic and endocrine coomplications , spread transfusion transmitted infections and formation of antibody (Ansari et al, 2022; Shah et al, 2019). These limitations have compelled researchers to search for novel therapeutic modalities (Fard et al., 2013; Ansari et al, 2022 ).

In recent years, induction of Fetal Hemoglobin (HbF) production pharmacologically is an promising treatment options for hemoglobinopathies (Fard et al., 2013; Thompson et al., 2018). Different HbF inducing agents like Hydroxyurea (HU), Butyrate derivatives, Azacitidine, Decitabine, Tricostatin-A are shown to be effective in decreasing clinical severity and complications of TDT (Fard et al., 2013). HU induces a 2-9 fold increase in γ-globin gene and being used for decades in thalassemia treatment (Jain et al., 2021; Fakredin et al., 2022). But its utility is limited due to its mild and ill sustained therapeutic effect in HbF synthesis (Green et al., 2016; Rigano et al.,2010). Thalidomide, an immunomodulatory drug also shown to produce significant and persistent rise in Hb in few small studies and several case reports (Aguilar-Lopez et al., 2008; Jain et al., 2021; Masera et al., 2010; Fakredin et al., 2022). It induces Gamma Globin gene expression by increasing reactive oxygen species-mediated p38 mitogen-activated protein kinase (MAPK) signaling and histone H4 acetylation (Aerbajinai et al., 2007).

Recent studies with combination of HU and Thalidomide have shown promising results in treatment of Thalassemia patients. However, most of those studies are retrospective or single arm nonrandomized trials (Shah et al., 2019) & The study population includes both adult and children age group (Ansari et al., 2022). So the effectiveness of combination therapy of Thalidomide and HU needs to be established in children through randomized trials.

So the goal of our study to evaluate the effectiveness of combination of Thalidomide and HU in comaprison to Thalisomide or HU alone in children with TDT through a three arm quasi randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as transfusion dependent thalassemia
* Age ranged from 3-18 years
* Blood transfusion more than 1 year.
* no bleeding disorder

Exclusion Criteria:

* Active systemic co-morbidity,
* Past personal or family history of thrombophilia,
* Recent fracture or recent major surgery
* Use of drugs that might affect Hb levels 15 days before enrollment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hb Level | 12 weeks after treatment initiation
  Change in Hb gm/dl after 3 month
Change in Blood transfusion frequency | 12 weeks after treatment initiation
  Change in Blood transfusion frequency after 3 month
Change in HbF | 12 weeks after treatment initiation
  Change in Hb F after 3 month

SECONDARY OUTCOMES:
Change in Biochemicals | 12 weeks after treatment initiation
  Change of S. Ferritin, SGPT, Creatinine, LDH, S. Bilirubin
Adverse effect | 12 weeks from treatment initiation
  Adverse effect of drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aerbajinai W, Zhu J, Gao Z, Chin K, Rodgers GP. Thalidomide induces gamma-globin gene expression through increased reactive oxygen species-mediated p38 MAPK signaling and histone H4 acetylation in adult erythropoiesis. Blood. 2007 Oct 15;110(8):2864-71. doi: 10.1182/blood-2007-01-065201. Epub 2007 Jul 9. PMID 17620452
- [Background] Aguilar-Lopez LB, Delgado-Lamas JL, Rubio-Jurado B, Perea FJ, Ibarra B. Thalidomide therapy in a patient with thalassemia major. Blood Cells Mol Dis. 2008 Jul-Aug;41(1):136-7. doi: 10.1016/j.bcmd.2008.03.001. Epub 2008 Apr 24. No abstract available. PMID 18439858
- [Background] Bou-Fakhredin R, De Franceschi L, Motta I, Cappellini MD, Taher AT. Pharmacological Induction of Fetal Hemoglobin in beta-Thalassemia and Sickle Cell Disease: An Updated Perspective. Pharmaceuticals (Basel). 2022 Jun 16;15(6):753. doi: 10.3390/ph15060753. PMID 35745672
- [Background] Cappellini MD, Porter JB, Viprakasit V, Taher AT. A paradigm shift on beta-thalassaemia treatment: How will we manage this old disease with new therapies? Blood Rev. 2018 Jul;32(4):300-311. doi: 10.1016/j.blre.2018.02.001. Epub 2018 Feb 12. PMID 29455932
- [Background] Chen JM, Zhu WJ, Liu J, Wang GZ, Chen XQ, Tan Y, Xu WW, Qu LW, Li JY, Yang HJ, Huang L, Cai N, Wang WD, Huang K, Xu JQ, Li GH, He S, Luo TY, Huang Y, Liu SH, Wu WQ, Lu QY, Zhou MG, Chen SY, Li RL, Hu ML, Huang Y, Wei JH, Li JM, Chen SJ, Zhou GB. Safety and efficacy of thalidomide in patients with transfusion-dependent beta-thalassemia: a randomized clinical trial. Signal Transduct Target Ther. 2021 Nov 18;6(1):405. doi: 10.1038/s41392-021-00811-0. PMID 34795208
- [Background] Costa E, Cappellini MD, Rivella S, Chilin A, Alessi E, Riccaboni M, Leufkens HGM, Luzzatto L. Emergent treatments for beta-thalassemia and orphan drug legislations. Drug Discov Today. 2022 Nov;27(11):103342. doi: 10.1016/j.drudis.2022.103342. Epub 2022 Sep 1. PMID 36058507
- [Background] Fard AD, Hosseini SA, Shahjahani M, Salari F, Jaseb K. Evaluation of Novel Fetal Hemoglobin Inducer Drugs in Treatment of beta-Hemoglobinopathy Disorders. Int J Hematol Oncol Stem Cell Res. 2013;7(3):47-54. PMID 24505535
- [Background] Farmakis D, Porter J, Taher A, Domenica Cappellini M, Angastiniotis M, Eleftheriou A. 2021 Thalassaemia International Federation Guidelines for the Management of Transfusion-dependent Thalassemia. Hemasphere. 2022 Jul 29;6(8):e732. doi: 10.1097/HS9.0000000000000732. eCollection 2022 Aug. PMID 35928543
- [Background] Fozza C, Pardini S, Giannico DB, Targhetta C, Di Tucci AA, Dessalvi P, Angelucci E, Dore F. Dramatic erythroid response to low-dose thalidomide in two patients with transfusion independent thalassemia and severe post-transfusional alloimmune hemolysis. Am J Hematol. 2015 Jul;90(7):E141. doi: 10.1002/ajh.24030. No abstract available. PMID 25850682
- [Background] Green NS, Manwani D, Qureshi M, Ireland K, Sinha A, Smaldone AM. Decreased fetal hemoglobin over time among youth with sickle cell disease on hydroxyurea is associated with higher urgent hospital use. Pediatr Blood Cancer. 2016 Dec;63(12):2146-2153. doi: 10.1002/pbc.26161. Epub 2016 Aug 30. PMID 27573582
- [Background] Hossain MS, Raheem E, Sultana TA, Ferdous S, Nahar N, Islam S, Arifuzzaman M, Razzaque MA, Alam R, Aziz S, Khatun H, Rahim A, Morshed M. Thalassemias in South Asia: clinical lessons learnt from Bangladesh. Orphanet J Rare Dis. 2017 May 18;12(1):93. doi: 10.1186/s13023-017-0643-z. PMID 28521805
- [Background] Jain M, Chakrabarti P, Dolai TK, Ghosh P, Mandal PK, Baul SN, De R. Comparison of efficacy and safety of thalidomide vs hydroxyurea in patients with Hb E-beta thalassemia - a pilot study from a tertiary care Centre of India. Blood Cells Mol Dis. 2021 May;88:102544. doi: 10.1016/j.bcmd.2021.102544. Epub 2021 Feb 3. PMID 33610115
- [Background] Li X, Hu S, Liu Y, Huang J, Hong W, Xu L, Xu H, Fang J. Efficacy of Thalidomide Treatment in Children With Transfusion Dependent beta-Thalassemia: A Retrospective Clinical Study. Front Pharmacol. 2021 Aug 12;12:722502. doi: 10.3389/fphar.2021.722502. eCollection 2021. PMID 34456732
- [Background] Masera N, Tavecchia L, Capra M, Cazzaniga G, Vimercati C, Pozzi L, Biondi A, Masera G. Optimal response to thalidomide in a patient with thalassaemia major resistant to conventional therapy. Blood Transfus. 2010 Jan;8(1):63-5. doi: 10.2450/2009.0102-09. No abstract available. PMID 20104280
- [Background] Rachmilewitz EA, Giardina PJ. How I treat thalassemia. Blood. 2011 Sep 29;118(13):3479-88. doi: 10.1182/blood-2010-08-300335. Epub 2011 Aug 2. PMID 21813448
- [Background] Rigano P, Pecoraro A, Calzolari R, Troia A, Acuto S, Renda D, Pantalone GR, Maggio A, Di Marzo R. Desensitization to hydroxycarbamide following long-term treatment of thalassaemia intermedia as observed in vivo and in primary erythroid cultures from treated patients. Br J Haematol. 2010 Dec;151(5):509-15. doi: 10.1111/j.1365-2141.2010.08397.x. Epub 2010 Oct 19. PMID 20955403
- [Background] Shah FT, Sayani F, Trompeter S, Drasar E, Piga A. Challenges of blood transfusions in beta-thalassemia. Blood Rev. 2019 Sep;37:100588. doi: 10.1016/j.blre.2019.100588. Epub 2019 Jul 6. PMID 31324412
- [Background] Taher A, Vichinsky E, Musallam K, Cappellini MD, Viprakasit V, authors. Weatherall D, editor. Guidelines for the Management of Non Transfusion Dependent Thalassaemia (NTDT) [Internet]. Nicosia (Cyprus): Thalassaemia International Federation; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK190453/ PMID 24672826
- [Background] Thompson AA, Walters MC, Kwiatkowski J, Rasko JEJ, Ribeil JA, Hongeng S, Magrin E, Schiller GJ, Payen E, Semeraro M, Moshous D, Lefrere F, Puy H, Bourget P, Magnani A, Caccavelli L, Diana JS, Suarez F, Monpoux F, Brousse V, Poirot C, Brouzes C, Meritet JF, Pondarre C, Beuzard Y, Chretien S, Lefebvre T, Teachey DT, Anurathapan U, Ho PJ, von Kalle C, Kletzel M, Vichinsky E, Soni S, Veres G, Negre O, Ross RW, Davidson D, Petrusich A, Sandler L, Asmal M, Hermine O, De Montalembert M, Hacein-Bey-Abina S, Blanche S, Leboulch P, Cavazzana M. Gene Therapy in Patients with Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2018 Apr 19;378(16):1479-1493. doi: 10.1056/NEJMoa1705342. PMID 29669226
- [Background] Weatherall DJ. The Evolving Spectrum of the Epidemiology of Thalassemia. Hematol Oncol Clin North Am. 2018 Apr;32(2):165-175. doi: 10.1016/j.hoc.2017.11.008. PMID 29458724
- [Background] Wolman IJ, Ortolani M. Some clinical features of Cooley's anemia patients as related to transfusion schedules. Ann N Y Acad Sci. 1969 Nov 20;165(1):407-14. doi: 10.1111/j.1749-6632.1969.tb27811.x. No abstract available. PMID 5260163
- [Background] Yassin AK. Promising Response to Thalidomide in Symptomatic beta-Thalassemia. Indian J Hematol Blood Transfus. 2020 Apr;36(2):337-341. doi: 10.1007/s12288-019-01231-5. Epub 2019 Nov 18. PMID 32425386